CLINICAL TRIAL: NCT00895583
Title: Planned Transition To Sirolimus-Based Therapy Versus Continued Tacrolimus-Based Therapy In Renal Allograft Recipients
Brief Title: Study Evaluating A Planned Transition From Tacrolimus To Sirolimus In Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0468E8-4500; B1741007
Record Dates: First submitted 2009-04-29; First posted 2009-05-08 (Estimated); Results first posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Graft Rejection; Kidney Transplant; Renal Allograft Recipients; Renal Transplant
Keywords: renal transplant; immunosuppression; sirolimus/rapamune; planned transition
MeSH Terms: interventions — Tacrolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I - Planned transition to sirolimus from tacrolimus (Experimental)
  Interventions: Drug: Tacrolimus; Drug: Sirolimus
- Group II - Continuation of tacrolimus (Active Comparator)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — During the screening phase, tacrolimus is provided by the investigator (not the Sponsor) and is dosed to achieve a target trough level determined by the investigator. Therefore, the dosage form, dosage, and frequency are determined by the investigator. Duration of treatment is from transplantation until randomization (from 90 to 150 days).
  Other Names: Prograf, Adagraf
  Arms: Group I - Planned transition to sirolimus from tacrolimus
Drug: Sirolimus — Following randomization, sirolimus is provided by the Sponsor in 1 and 2 mg oral tablets. Sirolimus is dosed once daily to achieve a target trough level of 7 to 15 ng/mL in the 1st year post-transplant and 5 - 15 ng/mL in the 2nd year post-transplant. Duration of treatment is from randomization through 2 years post-transplant (19 to 21 months).
  Other Names: Rapamune
  Arms: Group I - Planned transition to sirolimus from tacrolimus
Drug: Tacrolimus — During the study, tacrolimus is provided by the investigator (not the Sponsor) and is dosed to achieve a target trough level determined by the investigator. Therefore, the dosage form, dosage, and frequency are determined by the investigator. Duration of treatment is 2 years post-transplant.
  Other Names: Prograf, adagraf
  Arms: Group II - Continuation of tacrolimus

SUMMARY:
This study will look at the effect on long-term kidney function using tacrolimus right after a transplant and then switching to sirolimus at 3 to 5 months after the transplant.

ELIGIBILITY:
Inclusion Criteria:

At Screening:

* Male or female subjects aged 18 years or older.
* Recipients who are 14 days prior to transplantation up through 14 days after transplantation.
* Recipients of a primary, living- or deceased-donor renal allograft.
* All female and male subjects who are biologically capable of having children must agree and commit to the use of a reliable method of birth control for the duration of the study and for 3 months after the last dose of test article. A subject is biologically capable of having children even if he or she is using contraceptives or if his or her sexual partner is sterile or using contraceptives.

At Randomization:

* Ninety (90) to 150 days post-transplantation.
* Treatment with tacrolimus and an inosine monophosphate dehydrogenase (IMPDH) inhibitor initiated less than or equal to 30 days of transplantation and has remained on both for the 30 days prior to randomization.

Exclusion Criteria:

At Screening:

* Recipients of multiple organ transplants (i.e., any prior or concurrent transplantation of any organs including prior renal transplant. )
* Recipients of adult or pediatric en bloc kidney transplants.
* Recipients who required or will require desensitization protocols.
* Known history of focal segmental glomerulosclerosis (FSGS) or membranoproliferative glomerulonephritis (MPGN).
* Evidence of active systemic or localized major infection, as determined by the investigator.
* Received any investigational drugs or devices less than or equal to 30 days prior to transplantation.
* Known or suspected allergy to sirolimus (SRL), tacrolimus (TAC), inosine-monophosphate dehydrogenase (IMPDH) inhibitor, macrolide antibiotics, iothalamate, iodine, iodine-containing products, including contrast media other compounds related to these products/classes of medication, or shellfish.
* History of malignancy less than or equal to 3 years of screening (except for adequately treated basal cell or squamous cell carcinoma of the skin).
* Recipients who are known to be human immunodeficiency virus (HIV) positive.
* Women who are biologically capable of having children with a positive urine or serum pregnancy test at screening.
* Breastfeeding women.

At Randomization:

* Any major illness/condition that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in and completion of the study, or could preclude the evaluation of the subject's response.
* Planned treatment with immunosuppressive therapies other than those described in the protocol.
* Subjects who underwent corticosteroids withdrawal or avoidance and did not receive antibody induction at the time of transplantation with anti-thymocyte globulin (rabbit) (rATG) (Thymoglobulin®), anti-thymocyte globulin (equine) (Atgam®), or alemtuzumab (Campath®).
* Subjects who have had corticosteroid (CS) discontinued less than or equal to 30 days before randomization.
* Calculated glomerular filtration rate (GFR) less than 40 mL/min/1.73m2 using the simplified Modification of Diet in Renal Disease (MDRD) formula less than or equal to 2 weeks prior to randomization.
* Spot urine protein to creatinine ratio (UPr/Cr) greater than or equal to 0.5 less than or equal to 2 weeks prior to randomization.
* Banff (2007) grade 2 or higher acute T-cell-mediated or any acute antibody-mediated rejection at any time post-transplantation.
* Any acute rejection (biopsy-confirmed or presumed) less than or equal to 30 days before randomization.
* More than 1 episode of acute rejection (biopsy-confirmed or presumed).
* Known Banff (2007) interstitial fibrosis and tubular atrophy (IF/TA) greater than or equal to grade 2 or recurrent/de novo glomerular disease.
* Major surgery less than or equal to 2 weeks prior to randomization.
* Active post-operative complication, e.g. infection, delayed wound healing.
* Total white blood cell count less than 2,000/mm3 or absolute neutrophil count (ANC) less than 1000 or platelet count less than 100,000/mm3 less than or equal to 2 weeks prior to randomization.
* Fasting triglycerides greater than 400 mg/dL (greater than 4.5 mmol/L) or fasting total cholesterol greater than 300 mg/dL (greater than 7.8 mmol/L) less than or equal to 2 weeks prior to randomization regardless of whether or not on lipid-lowering therapy.
* Women who are biologically capable of having children with a positive urine or serum pregnancy test at randomization.
* Breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2009-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (22):
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Portland, Maine
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
- Pfizer Investigational Site, Ciudad de Buenos Aires, Buenos Aires, Argentina
- Australia (3):
  - Pfizer Investigational Site, Randwick, New South Wales
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Nedlands, Western Australia
- Brazil (3):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Bela Vista, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, Berlin, Germany
- Italy (2):
  - Pfizer Investigational Site, Milan, Milano
  - Pfizer Investigational Site, Milan
- Spain (6):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Santander

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus: Participants received tacrolimus (extended-release formulation not permitted) within 30 days of transplant, dosed according to center's standard of care. At 3-5 months post-transplant, participants were randomized, tacrolimus was discontinued (withdrawal was to be completed within 2 weeks [maximum of 4 weeks] of sirolimus initiation) and participants received sirolimus tablets, orally, at a dose to achieve trough levels of 7-15 nanograms per milliliter (ng/mL) during the first year post-transplant, then 5-15 ng/mL. Participants remained on an inosine monophosphate dehydrogenase (IMPDH) inhibitor (mycophenolate mofetil [MMF] or mycophenolate sodium [MPS]; switching between the two was permitted). Corticosteroids were maintained at a minimum of 2.5 milligrams per day (mg/day) of prednisone (or equivalent); withdrawal was prohibited after randomization. Participants received study drug during the post-randomization period for up to a maximum of 18 months post-transplant.
- Tacrolimus: Participants received tacrolimus (extended-release formulation not permitted) within 30 days of transplant, dosed according to center's standard of care. At 3-5 months post-transplant, participants were randomized and tacrolimus continued. Participants remained on an IMPDH inhibitor (MMF or MPS; switching between the two was permitted). Corticosteroids were maintained at a minimum of 2.5 mg/day of prednisone (or equivalent); withdrawal was prohibited after randomization. Participants received study drug during the post-randomization period for up to a maximum of 18 months post-transplant.
Period: Overall Study
Arm/Group | Sirolimus | Tacrolimus
Started | 131 | 123
Completed | 87 | 111
Not Completed | 44 | 12
Not completed — Adverse Event | 28 | 4
Not completed — Death | 2 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lack of Efficacy | 5 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: all randomized participants who received at least one dose of the assigned therapy after randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus | Tacrolimus | Total
Number analyzed (Participants) | 131 | 123 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (13.03) | 52.4 (12.05) | 51.5 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 46 | 88
  Male | 89 | 77 | 166

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Improvement of Greater Than or Equal to [≥]5 Milliliters Per Minute Per 1.73 Square Meters (mL/Min/m^2) in Calculated Glomerular Filtration Rate (GFR) at 24 Months Post-Transplantation (On-Therapy Analysis)
Description: GFR was calculated using the Modified Diet in Renal Disease (MDRD) equation using either serum creatinine traceable to isotope dilution mass spectrometry (IDMS) or serum creatinine not traceable to IDMS.
Time Frame: Baseline, Month 24
Population: On-Therapy Population (24 Months): all randomized participants who remained on assigned study therapy through 24 months post-transplantation.
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 86 | 109
percentage of participants | 33.7 | 42.2
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.239, Fisher Exact — Two-sided alpha equals (=) 0.05; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.4 to 1.3]

2. Secondary Outcome: Percentage of Participants With Improvement of ≥5 mL/Min/m^2 in Calculated GFR at 12 Months Post-Transplantation (On-Therapy Analysis)
Description: GFR was calculated using the MDRD equation using either serum creatinine traceable to IDMS or serum creatinine not traceable to IDMS.
Time Frame: Baseline, Month 12
Population: On-Therapy Population (12 Months): all randomized participants who remained on assigned study therapy through 12 months post-transplantation.
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 109 | 116
percentage of participants | 39.4 | 44.8
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.422, Fisher Exact — Alpha was unadjusted; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.5 to 1.4]

3. Secondary Outcome: Percentage of Participants With Improvement of ≥5 mL/Min/m^2 in Calculated GFR at 12 and 24 Months Post-Transplantation (Intent-to-Treat [ITT] Analysis)
Description: as for outcome 2
Time Frame: Baseline, Months 12 and 24
Population: ITT Population: all randomized participants who received at least 1 dose of the assigned therapy after randomization. Missing GFR was imputed as follows: 1) GFR equals (=)0 after graft loss and 2) last observed value prior to missing was carried forward for death (with functioning graft), early termination or skipped assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants
  Month 12 | 38.2 | 42.3
  Month 24 | 33.6 | 40.7
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Month 12; Test type: Superiority or Other; p = 0.524, Fisher Exact — Alpha was unadjusted; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.5 to 1.4]
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Month 24; Test type: Superiority or Other; p = 0.298, Fisher Exact — Alpha was unadjusted; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.4 to 1.2]

4. Secondary Outcome: Percentage of Participants With Improvement of ≥7.5 mL/Min/m^2 in Calculated GFR at 12 and 24 Months Post-Transplantation
Description: as for outcome 2
Time Frame: Baseline, Months 12 and 24
Population: ITT Population. Missing GFR was imputed as follows: 1) GFR=0 after graft loss and 2) last observed value prior to missing was carried forward for death (with functioning graft), early termination or skipped assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants
  Month 12 | 24.4 | 35.8
  Month 24 | 25.2 | 30.9
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Month 12; Test type: Superiority or Other; p = 0.055, Fisher Exact — Alpha was unadjusted; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.3 to 1.0]
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Month 24; Test type: Superiority or Other; p = 0.330, Fisher Exact — Alpha was unadjusted; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.4 to 1.3]

5. Secondary Outcome: Percentage of Participants With Improvement of ≥10 mL/Min/m^2 in Calculated GFR at 12 and 24 Months Post-Transplantation
Description: as for outcome 2
Time Frame: Baseline, Months 12 and 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants
  Month 12 | 19.8 | 23.6
  Month 24 | 22.1 | 22.0
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Month 12; Test type: Superiority or Other; p = 0.543, Fisher Exact — Alpha was unadjusted; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.4 to 1.5]
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Month 24; Test type: Superiority or Other; p = 1.000, Fisher Exact — Alpha was unadjusted; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.6 to 1.8]

6. Secondary Outcome: Calculated GFR Using MDRD (On-Therapy Analysis)
Description: GFR was calculated using the MDRD equation using either serum creatinine traceable to IDMS or serum creatinine not traceable to IDMS. Baseline was defined as the last nonmissing assessment before or on the date of the first dose of test article.
Time Frame: Baseline, Months 6, 12, 18, and 24
Population: On-Therapy Population: all participants who remained on assigned study therapy up to the point of discontinuation. number (n)=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
mL/min/1.73 m^2
  Baseline (n=131,123) | 58.5 (14.3) | 57.4 (14.1)
  Month 6 (n=125,120) | 61.6 (14.9) | 57.6 (14.2)
  Month 12 (n=109,116) | 59.6 (16.4) | 61.3 (14.3)
  Month 18 (n=99,111) | 60.0 (15.0) | 59.8 (17.1)
  Month 24 (n=86,109) | 59.4 (18.0) | 58.4 (14.9)

7. Secondary Outcome: Change From Randomization in Calculated GFR Using MDRD (On-Therapy Analysis)
Description: as for outcome 6
Time Frame: Baseline, Months 6, 12, 18, and 24
Population: On-Therapy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
mL/min/1.73 m^2
  Month 6 (n=125,120) | 2.7 (1.1) | 0.0 (0.8)
  Month 12 (n=109,116) | 1.5 (1.2) | 3.4 (1.1)
  Month 18 (n=99,111) | 2.2 (1.2) | 1.5 (1.3)
  Month 24 (n=86,109) | 1.2 (1.6) | 0.6 (1.3)
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Change from randomization at Month 6; Test type: Superiority or Other; p = 0.019, ANCOVA — Alpha was unadjusted; Analysis of covariance (ANCOVA) with treatment as a factor and baseline GFR as a covariate; Least Squares (LS) Mean Difference = 3.0, 95% CI 2-sided [0.5 to 5.5], Standard Error of Mean 1.3
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Change from randomization at Month 12; Test type: Superiority or Other; p = 0.215, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline GFR as a covariate; LS Mean Difference = -1.9, 95% CI 2-sided [-4.8 to 1.1], Standard Error of Mean 1.5
Statistical Analysis 3: Comparison: Sirolimus vs Tacrolimus; Change from randomization at Month 18; Test type: Superiority or Other; p = 0.722, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline GFR as a covariate; LS Mean Difference = 0.6, 95% CI 2-sided [-2.7 to 3.9], Standard Error of Mean 1.7
Statistical Analysis 4: Comparison: Sirolimus vs Tacrolimus; Change from randomization at Month 24; Test type: Superiority or Other; p = 0.710, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline GFR as a covariate; LS Mean Difference = 0.7, 95% CI 2-sided [-3.0 to 4.4], Standard Error of Mean 1.9

8. Secondary Outcome: Slope of Calculated GFR (MDRD) From Randomization to 24 Months Post-Transplantation (On-Therapy Analysis)
Description: GFR was calculated using the MDRD equation using either serum creatinine traceable to IDMS or serum creatinine not traceable to IDMS. Timepoints were calculated as study days, relative to the time of randomization of study medication. All available on-therapy values were included. Observed data were multiplied by a scale factor of 365, expressing the slope as an annual change.
Time Frame: Baseline, Month 24
Population: On-Therapy analysis of the slope comprised the data collected from the on-therapy evaluations for all the participants in the ITT population; data collected from participants receiving sirolimus during the first 3 weeks post-randomization for safety monitoring were excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73 m^2 per year
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
mL/min/1.73 m^2 per year | -0.9 [-2.7 to 0.8] | 0.9 [-0.7 to 2.5]
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Slope difference (sirolimus [SRL] minus tacrolimus [TAC]); Test type: Superiority or Other; p = 0.131, Random coefficient model; Slope difference (SRL-TAC) = -1.8, 95% CI 2-sided [-4.2 to 0.5] — Random coefficient model with GFR as the dependent variable and study day as the independent variable

9. Secondary Outcome: Serum Creatinine (On-Therapy Analysis)
Description: Serum creatinine was measured in micromillimoles per liter (mcmol/L). Baseline was defined as the last nonmissing assessment before or on the date of the first dose of test article.
Time Frame: Baseline, Months 6, 12, 18, and 24
Population: On-Therapy Population: all participants who remained on assigned study therapy up to the point of discontinuation. n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
mcmol/L
  Baseline (n=131,123) | 118.3 (24.8) | 117.7 (27.9)
  Month 6 (n=125,120) | 113.9 (27.6) | 117.0 (28.2)
  Month 12 (n=109,116) | 119.6 (37.5) | 109.4 (24.6)
  Month 18 (n=99,111) | 116.9 (33.1) | 114.2 (30.4)
  Month 24 (n=86,109) | 122.9 (48.8) | 117.5 (42.8)

10. Secondary Outcome: Change From Randomization in Serum Creatinine (On-Therapy Analysis)
Description: Serum creatinine was measured in mcmol/L. Baseline was defined as the last assessment prior to first administration of study drug.
Time Frame: Baseline, Months 6, 12, 18, and 24
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mcmol/L
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
mcmol/L
  Month 6 (n=125,120) | -4.1 (2.0) | -0.0 (1.4)
  Month 12 (n=109,116) | -0.3 (2.9) | -7.0 (1.9)
  Month 18 (n=99,111) | -3.0 (2.5) | -1.9 (2.3)
  Month 24 (n=86,109) | 3.2 (4.6) | 0.5 (3.7)
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Change from randomization at Month 6; Test type: Superiority or Other; p = 0.105, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline serum creatinine as a covariate; LS Mean Difference = -3.9, 95% CI 2-sided [-8.6 to 0.8], Standard Error of Mean 2.4
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Change from randomization at Month 12; Test type: Superiority or Other; p = 0.023, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline serum creatinine as a covariate; LS Mean Difference = 7.7, 95% CI 2-sided [1.1 to 14.3], Standard Error of Mean 3.3
Statistical Analysis 3: Comparison: Sirolimus vs Tacrolimus; Change from randomization at Month 18; Test type: Superiority or Other; p = 0.955, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline serum creatinine as a covariate; LS Mean Difference = -0.2, 95% CI 2-sided [-6.8 to 6.4], Standard Error of Mean 3.4
Statistical Analysis 4: Comparison: Sirolimus vs Tacrolimus; Change from randomization at Month 24; Test type: Superiority or Other; p = 0.582, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline serum creatinine as a covariate; LS Mean Difference = 3.2, 95% CI 2-sided [-8.2 to 14.6], Standard Error of Mean 5.8

11. Secondary Outcome: Percentage of Participants With Biopsy-Confirmed Acute Rejection (BCAR), Graft Loss, or Death From Randomization to 24 Months Post-Transplantation
Description: Biopsy-confirmed acute rejection was defined according to updated Banff criteria (2007) for renal allograft rejection. Graft loss was defined as physical loss (nephrectomy or retransplantation), functional loss (requiring dialysis for greater than or equal to [≥]56 days with no return of graft function), or death.
Time Frame: Post-randomization to Month 24 post-transplantation
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants | 11.5 | 2.4
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.006, Fisher Exact — Alpha was unadjusted

12. Secondary Outcome: Percentage of Participants With Graft Loss (Including Death) at 12 and 24 Months Post-Randomization
Description: Graft loss was defined as physical loss (nephrectomy or retransplantation), functional loss (requiring dialysis for ≥56 days with no return of graft function), or death.
Time Frame: Post-randomization to Months 12 and 24 Post-Transplantation
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants
  Month 12 | 0.8 | 0.0
  Month 24 | 3.8 | 0.8
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Post-randomization to Month 12 Post-transplantation; Test type: Superiority or Other; p = 1.000, Fisher Exact — Alpha was unadjusted
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Post-randomization to Month 24 post-transplantation; Test type: Superiority or Other; p = 0.215, Fisher Exact — Alpha was unadjusted

13. Secondary Outcome: Percentage of Participants With BCAR Post-Randomization to 6, 12, 18, and 24 Months Post-Transplantation
Description: BCAR was defined according to updated Banff criteria (2007) for renal allograft rejection.
Time Frame: Post-Randomization to 6, 12, 18, and 24 months Post-Transplantation
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants
  Month 6 | 1.5 | 0.0
  Month 12 | 5.3 | 0.8
  Month 18 | 6.9 | 1.6
  Month 24 | 8.4 | 1.6
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Month 6; Test type: Superiority or Other; p = 0.499, Fisher Exact — Alpha was unadjusted
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Month 12; Test type: Superiority or Other; p = 0.067, Fisher Exact — Alpha was unadjusted
Statistical Analysis 3: Comparison: Sirolimus vs Tacrolimus; Month 18; Test type: Superiority or Other; p = 0.061, Fisher Exact — Alpha was unadjusted
Statistical Analysis 4: Comparison: Sirolimus vs Tacrolimus; Month 24; Test type: Superiority or Other; p = 0.020, Fisher Exact — Alpha was unadjusted

14. Secondary Outcome: Percentage of Participants With First On-Therapy BCAR From Transplantation Occurring at 12 and 24 Months
Description: Defined as the first BCAR occurring during the On-Therapy period based on the ITT population. Time to first BCAR was the days from transplantation to the date of BCAR.
Time Frame: Months 12 and 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants
  Month 12 | 5.1 | 0.0
  Month 24 | 9.3 | 0.9

15. Secondary Outcome: Number of Participants With BCAR by Severity of First BCAR and Time of Onset From Post-Randomization to 6, 12, 18, and 24 Months Post-Transplant
Description: BCAR was categorized as antibody-mediated (AM) or T-cell. AM BCAR severity was graded as Grade I (mild), Grade II (moderate), and Grade III (severe). T-cell BCAR severity was graded as 'Grade Ia, Ib (mild), Grade IIa, IIb (moderate), and Grade III (severe). If a participant had both T-cell BCAR and antibody-mediated BCAR on the first rejection, the participant was counted in each category.
Time Frame: Months 6, 12, 18, and 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
participants
  Month 6, AM Grade I | 0 | 0
  Month 6, AM Grade II | 0 | 0
  Month 6, AM Grade III | 0 | 0
  Month 6, T-cell Grade Ia, Ib | 2 | 0
  Month 6, T-cell Grade IIa, IIb | 0 | 0
  Month 6, T-cell Grade III | 0 | 0
  Month 12, AM Grade I | 1 | 0
  Month 12, AM Grade II | 0 | 0
  Month 12, AM Grade III | 1 | 0
  Month 12, T-cell Grade Ia, Ib | 5 | 0
  Month 12, T-cell Grade IIa, IIb | 1 | 1
  Month 12, T-cell Grade III | 0 | 0
  Month 18, AM Grade I | 1 | 1
  Month 18, AM Grade II | 0 | 0
  Month 18, AM Grade III | 1 | 0
  Month 18, T-cell Grade Ia, Ib | 7 | 1
  Month 18, T-cell Grade IIa, IIb | 1 | 1
  Month 18, T-cell Grade III | 0 | 0
  Month 24, AM Grade I | 2 | 1
  Month 24, AM Grade II | 1 | 0
  Month 24, AM Grade III | 1 | 0
  Month 24, T-cell Grade Ia, Ib | 8 | 1
  Month 24, T-cell Grade IIa, IIb | 1 | 1
  Month 24, T-cell Grade III | 0 | 0

16. Secondary Outcome: Percentage of Participants With Antibody Use in Treatment of Acute Rejection
Description: Number of participants who experienced an adverse event (AE) of rejection was used as the denominator in the determination of percentage of participants with antibody use in treatment of acute rejection.
Time Frame: On Therapy Period (up to 21 months post-randomization) and Off-Therapy Period (up to 24 months post-transplantation)
Population: Safety Population; only participants with an AE of rejection were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 15 | 4
percentage of participants
  On-therapy Period | 60.0 | 75.0
  Off-therapy Period | 40.0 | 25.0
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; On-therapy Period; Test type: Superiority or Other; p = 1.000, Fisher Exact — Alpha was unadjusted
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Off-therapy Period; Test type: Superiority or Other; p = 1.000, Fisher Exact — Alpha was unadjusted

17. Secondary Outcome: Percentage of Participants With Anemia, Thrombocytopenia, or Leukopenia
Description: Anemia was defined as hemoglobin less than or equal to (≤)10 grams per deciliter (g/dL); leukopenia was defined as white blood cell (WBC) count ≤2000 per cubic millimeters (/mm^3); and thrombocytopenia was defined as platelets ≤100,000/mm^3. Baseline was defined as the last nonmissing assessment before or on the date of the first dose of test article.
Time Frame: Baseline, Months 12 and 24
Population: Safety Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 122
percentage of participants
  Baseline (n=131,122) | 4.6 | 1.6
  Month 12 (n=110,116) | 9.1 | 2.6
  Month 24 (n=89,112) | 3.4 | 4.5
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Baseline; Test type: Superiority or Other; p = 0.284, Fisher Exact — Alpha was unadjusted
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Month 12; Test type: Superiority or Other; p = 0.046, Fisher Exact — Alpha was unadjusted
Statistical Analysis 3: Comparison: Sirolimus vs Tacrolimus; Month 24; Test type: Superiority or Other; p = 1.000, Fisher Exact — Alpha was unadjusted

18. Secondary Outcome: Change From Baseline (Pre-Randomization) to 12 and 24 Months Post-Transplantation in Fasting Lipid Parameters (Millimoles Per Liter [mmol/L])
Description: Parameters assessed included total cholesterol (TC), triglycerides, low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C); collected when participant was in a fasting state.
Time Frame: Baseline, Months 12 and 24
Population: Safety Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 96 | 107
mmol/L
  TC, Change at Month 12 (n=96,107) | 0.66 (0.10) | -0.12 (0.07)
  TC, Change at Month 24 (n=74,88) | 0.51 (0.14) | -0.08 (0.09)
  HDL-C, Change at Month 12 (n=90,99) | -0.00 (0.03) | 0.01 (0.02)
  HDL-C, Change at Month 24 (n=69,81) | 0.01 (0.04) | 0.01 (0.03)
  LDL-C, Change at Month 12 (n=87,98) | 0.43 (0.09) | -0.06 (0.07)
  LDL-C, Change at Month 24 (n=66,78) | 0.34 (0.13) | -0.06 (0.08)
  Triglycerides, Change at Month 12 (n=94,104) | 0.47 (0.11) | -0.18 (0.07)
  Triglycerides, Change at Month 24 (n=73,86) | 0.43 (0.10) | 0.07 (0.12)
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; TC, Month 12; Test type: Superiority or Other; p < 0.001, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.81, Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; TC, Month 24; Test type: Superiority or Other; p < 0.001, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Mean = 0.61, Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Sirolimus vs Tacrolimus; HDL-C, Month 12; Test type: Superiority or Other; p = 0.824, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = -0.01, Standard Error of Mean 0.03
Statistical Analysis 4: Comparison: Sirolimus vs Tacrolimus; HDL-C, Month 24; Test type: Superiority or Other; p = 0.735, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = -0.02, Standard Error of Mean 0.05
Statistical Analysis 5: Comparison: Sirolimus vs Tacrolimus; LDL-C, Month 12; Test type: Superiority or Other; p < 0.001, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.49, Standard Error of Mean 0.11
Statistical Analysis 6: Comparison: Sirolimus vs Tacrolimus; LDL-C, Month 24; Test type: Superiority or Other; p = 0.001, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.42, Standard Error of Mean 0.13
Statistical Analysis 7: Comparison: Sirolimus vs Tacrolimus; Triglycerides, Month 12; Test type: Superiority or Other; p < 0.001, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.65, Standard Error of Mean 0.13
Statistical Analysis 8: Comparison: Sirolimus vs Tacrolimus; Triglycerides, Month 24; Test type: Superiority or Other; p = 0.028, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.37, Standard Error of Mean 0.16

19. Secondary Outcome: Percentage of Participants Requiring Anti-Hypertensive Medication, Diabetes Agents, Lipid-Lowering Agents, or Erythropoiesis Stimuating Agents (ESAs)
Time Frame: Baseline, Months 12 and 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants
  Baseline, Anti-hypertensives | 95.4 | 92.7
  Month 12, Anti-hypertensives | 75.6 | 69.9
  Month 24, Anti-hypertensives | 61.8 | 65.9
  Baseline, Diabetes agents (insulin) | 46.6 | 47.2
  Month 12, Diabetes agents (insulin) | 26.0 | 26.0
  Month 24, Diabetes agents (insulin) | 18.3 | 25.2
  Baseline, Diabetes agents (non-insulin) | 14.5 | 17.9
  Month 12, Diabetes agents (non-insulin) | 10.7 | 13.8
  Month 24, Diabetes agents (non-insulin) | 9.2 | 13.0
  Baseline, Lipid-lowering agents | 46.6 | 60.2
  Month 12, Lipid-lowering agents | 55.7 | 54.5
  Month 24, Lipid-lowering agents | 47.3 | 49.6
  Baseline, ESAs | 50.4 | 43.1
  Month 12, ESAs | 7.6 | 2.4
  Month 24, ESAs | 3.8 | 2.4
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Anti-hypertensives, Baseline; Test type: Superiority or Other; p = 0.429, Fisher Exact — Alpha was unadjusted
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Anti-hypertensives, Month 12; Test type: Superiority or Other; p = 0.326, Fisher Exact — Alpha was unadjusted
Statistical Analysis 3: Comparison: Sirolimus vs Tacrolimus; Anti-hypertensives, Month 24; Test type: Superiority or Other; p = 0.517, Fisher Exact — Alpha was unadjusted
Statistical Analysis 4: Comparison: Sirolimus vs Tacrolimus; Diabetes agents (insulin), Baseline; Test type: Superiority or Other; p = 1.000, Fisher Exact — Alpha was unadjusted
Statistical Analysis 5: Comparison: Sirolimus vs Tacrolimus; Diabetes agent (insulin), Month 12; Test type: Superiority or Other; p = 1.000, Fisher Exact — Alpha was unadjusted
Statistical Analysis 6: Comparison: Sirolimus vs Tacrolimus; Diabetes agent (insulin), Month 24; Test type: Superiority or Other; p = 0.223, Fisher Exact — Alpha was unadjusted
Statistical Analysis 7: Comparison: Sirolimus vs Tacrolimus; Diabetes agent (non-insulin), Baseline; Test type: Superiority or Other; p = 0.498, Fisher Exact — Alpha was unadjusted
Statistical Analysis 8: Comparison: Sirolimus vs Tacrolimus; Diabetes agent (non-insulin), Month 12; Test type: Superiority or Other; p = 0.566, Fisher Exact — Alpha was unadjusted
Statistical Analysis 9: Comparison: Sirolimus vs Tacrolimus; Diabetes agent (non-insulin), Month 24; Test type: Superiority or Other; p = 0.423, Fisher Exact — Alpha was unadjusted
Statistical Analysis 10: Comparison: Sirolimus vs Tacrolimus; Lipid-lowering agents, Baseline; Test type: Superiority or Other; p = 0.033, Fisher Exact — Alpha was unadjusted
Statistical Analysis 11: Comparison: Sirolimus vs Tacrolimus; Lipid-lowering agents, Month 12; Test type: Superiority or Other; p = 0.900, Fisher Exact — Alpha was unadjusted
Statistical Analysis 12: Comparison: Sirolimus vs Tacrolimus; Lipid-lowering agents, Month 24; Test type: Superiority or Other; p = 0.802, Fisher Exact — Alpha was unadjusted
Statistical Analysis 13: Comparison: Sirolimus vs Tacrolimus; ESAs, Baseline; Test type: Superiority or Other; p = 0.260, Fisher Exact — Alpha was unadjusted
Statistical Analysis 14: Comparison: Sirolimus vs Tacrolimus; ESAs, Month 12; Test type: Superiority or Other; p = 0.086, Fisher Exact — Alpha was unadjusted
Statistical Analysis 15: Comparison: Sirolimus vs Tacrolimus; ESAs, Month 24; Test type: Superiority or Other; p = 0.723, Fisher Exact — Alpha was unadjusted

20. Secondary Outcome: Spot and 24 Hour Urine Protein to Creatinine Ratio (UPr/Cr)
Description: Baseline was defined as the last nonmissing assessment before or on the date of the first dose of test article.
Time Frame: Baseline and Months 12 and 24
Population: Safety Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: UPr/Cr
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 127 | 120
UPr/Cr
  Baseline (n=127,120) | 0.180 (0.1413) | 0.195 (0.1477)
  Month 12 (n=112,108) | 0.353 (0.3677) | 0.208 (0.2234)
  Month 24 (n=102,106) | 0.510 (0.7887) | 0.300 (0.6154)
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Change from pre-randomization at Month 12; treatment ratio (SRC/TAC) in adjusted geometric mean fold-change from baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — Alpha was unadjusted; ANCOVA model with change in the logarithmic Upr/Cr as dependent variable, treatment and logarithmic pre-randomization value as covariate; Treatment Ratio = 1.71, 95% CI 2-sided [1.38 to 2.11]
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Change from pre-randomization at Month 24; treatment ratio (SRC/TAC) in adjusted geometric mean fold-change from baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — Alpha was unadjusted; [statistical method as in outcome 20, analysis 1]; Treatment Ratio = 1.77, 95% CI 2-sided [1.39 to 2.26]

21. Secondary Outcome: Percentage of Participants With Angiotensin Converting Enzyme Inhibitor (ACEI) or Angiotensin II Receptor Block (ARB) Use
Description: Included ACEI or ARB use prior to randomization, during the on-therapy period (up to 19 to 21 months post randomization) and the off-therapy period (up to 24 months post-transplantation).
Time Frame: Pre-randomization, On-Therapy Period (up to 21 months post-randomization), and Off-Therapy Period (up to 24 months post-transplantation)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants
  Pre-randomization | 46.6 | 46.3
  On-Therapy Period | 43.5 | 29.3
  Off-Therapy Period | 32.1 | 18.7
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Pre-randomization; Test type: Superiority or Other; p = 1.000, Fisher Exact — Alpha was unadjusted
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; On-Therapy Period; Test type: Superiority or Other; p = 0.020, Fisher Exact — Alpha was unadjusted
Statistical Analysis 3: Comparison: Sirolimus vs Tacrolimus; Off-Therapy Period; Test type: Superiority or Other; p = 0.021, Fisher Exact — Alpha was unadjusted

22. Secondary Outcome: Percentage of Participants With Stomatitis
Description: Includes adverse events based on categorization by the investigator as stomatitis, regardless of the event preferred term in Medical Dictionary for Regulatory Activities (MedDRA)
Time Frame: From randomization up to 24 months after transplantation (On-Therapy)
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants | 28.2 | 1.6
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p < 0.001, Fisher Exact — Alpha is unadjusted

23. Secondary Outcome: Percentage of Participants Requiring Treatment for Stomatitis by Treatment Type
Description: Included treatments (analgesics, dental paste, topical antifungal, topical steroids, or other) prior to randomization, during the on-therapy period (up to 19 to 21 months post-randomization) and the off-therapy period (up to 24 months post-transplantation).
Time Frame: On-Therapy Period (up to 21 months post-randomization) and Off-Therapy Period (up to 24 months post-transplantation)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants
  On-Therapy Period, any treatment | 17.6 | 2.4
  Off-Therapy Period, any treatment | 3.1 | 1.6
  On-Therapy, analgesics | 0.8 | 0.0
  On-Therapy, dental paste | 3.8 | 0.8
  On-Therapy, topical steroids | 5.3 | 0.0
  On-Therapy, other | 10.7 | 2.4
  Off-Therapy, topical steroids | 1.5 | 0.0
  Off-Therapy, other | 1.5 | 1.6
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; On-Therapy Period, any treatment; Test type: Superiority or Other; p < 0.001, Fisher Exact — Alpha was unadjusted
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Off-Therapy Period, any treatment; Test type: Superiority or Other; p = 0.685, Fisher Exact — Alpha was unadjusted

24. Secondary Outcome: Change From Pre-Randomization to 12 Months Post-Transplantation in Hemoglobin A1C (Liter Per Liter [L/L])
Description: Ratio of hemoglobin A1c to normal hemoglobin.
Time Frame: Baseline, Month 12
Population: Safety Population
Measure: Mean (Standard Error); unit: L/L
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 86 | 98
L/L | -0.00 (0.00) | 0.00 (0.00)
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.521, ANCOVA — Alpha was unadjusted; Difference in Adjusted Means = -0.00, Standard Error of Mean 0.00

25. Secondary Outcome: Change From Pre-Randomization to 12 Months Post-Transplantation in Fasting Glucose (mmol/L)
Time Frame: Baseline, Month 12
Population: Safety Population
Measure: Mean (Standard Error); unit: mmol
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 101 | 112
mmol | -0.50 (0.31) | -0.23 (0.20)
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.265, ANCOVA — Alpha is unadjusted; Difference in Adjusted Means = -0.28, Standard Error of Mean 0.25 — ANCOVA with treatment as a factor and baseline as a covariate

26. Secondary Outcome: Change From Pre-Randomization to 12 Months Post-Transplantation in Fasting Insulin (Picomoles Per Liter [Pmol/L])
Time Frame: Baseline, Month 12
Population: Safety Population
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 71 | 84
pmol/L | 27.25 (21.97) | 17.14 (11.85)
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.672, ANCOVA — Alpha was unadjusted; Difference in Adjusted Means = 10.02, Standard Error of Mean 23.61 — ANCOVA with treatment as a factor and baseline as a covariate

27. Secondary Outcome: Change From Pre-Randomization to 12 Months Post-Transplantation in Weight (Kilograms [kg])
Time Frame: Baseline, Month 12
Population: Safety Population
Measure: Mean (Standard Error); unit: kg
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 104 | 113
kg | 1.61 (0.51) | 2.03 (0.44)
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.504, ANCOVA — Alpha was unadjusted; Difference in Adjusted Means = -0.45, Standard Error of Mean 0.67 — ANCOVA with treatment as a factor and baseline as a covariate

28. Secondary Outcome: Change From Pre-Randomization to 12 Months Post-Transplantation in Waist Circumference(Centimeters [cm])
Time Frame: Baseline, Month 12
Population: Safety Population
Measure: Mean (Standard Error); unit: cm
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 98 | 105
cm | 1.13 (0.73) | 2.21 (1.00)
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.637, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = -0.56, Standard Error of Mean 1.18

29. Secondary Outcome: Change From Pre-Randomization to 12 Months Post-Transplantation in Homeostasis Model Assessment Insulin Resistance (HOMA-IR; Fasting)
Description: The HOMA-IR measures insulin resistance based on fasting glucose and insulin measurements:
  HOMA-IR = fasting plasma glucose (mmol/L) multiplied by (*) fasting plasma insulin in microunits per liter (µU/L) divided by (/) 22.5.
  Participants taking insulin within 12 hours were excluded from the analysis.
Time Frame: Baseline, Month 12
Population: Safety Population
Measure: Mean (Standard Error); unit: insulin resistance score
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 66 | 77
insulin resistance score | 1.14 (1.37) | 1.10 (0.70)
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.955, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.08, Standard Error of Mean 1.48

30. Secondary Outcome: Change From Pre-Randomization to 12 Months Post-Transplantation in HOMA-Beta Cell (HOMA-B; Fasting)
Description: The Homeostasis Model Assessment (HOMA) estimates steady state beta cell function (%B) as a percentage of a normal reference population.
  HOMA-B = 20 * insulin (µU/L) / fasting plasma glucose (mmol/L) minus (-) 3.5 Participants taking insulin within 12 hours were excluded from the analysis.
Time Frame: Baseline, Month 12
Population: Safety Population
Measure: Mean (Standard Error); unit: percentage beta cell function
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 66 | 77
percentage beta cell function | 230.23 (214.68) | 26.05 (21.99)
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.279, ANCOVA — Alpha was unadjusted; ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 216.29, Standard Error of Mean 198.84

31. Secondary Outcome: Change From Pre-Randomization to 12 Months Post-Transplantation in Body Mass Index (BMI; in Kilograms Per Square Meter [kg/m^2])
Description: BMI = Weight (kg)/(Height*Height) (square meters [m^2]).
Time Frame: Baseline, Month 12
Population: Safety Population
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 101 | 109
kg/m^2 | 0.53 (0.18) | 0.75 (0.15)
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.337, ANCOVA — Alpha was unadjusted; Difference in Adjusted Means = -0.22, Standard Error of Mean 0.23

32. Secondary Outcome: Percentage of Participants With New-Onset Diabetes
Description: Participants were considered as having new onset diabetes during the On-therapy period if any of the below events emerged from baseline to Month 24: 1) at least 30 days continuous, or at least 25 days non-stop (without gap) use of any diabetic treatment after randomization; 2) a fasting glucose greater than or equal to (≥)126 milligrams per deciliter (mg/dL) after randomization; or 3) a non-fasting glucose ≥200 mg/dL after randomization, were included in the new-onset diabetes population. Events at Months 12 or 24 occurred from baseline to On-therapy Month 12 and from On-therapy Months 12 to 24, respectively.
Time Frame: From Baseline to On-Therapy Month 12, from Baseline to On-Therapy Month 24, and from On-Therapy Month 12 up to On-Therapy Month 24
Population: Safety Population; participants at risk of new-onset diabetes mellitus at the beginning of the analysis interval were included and those with pre-existing diabetes were excluded from the analysis. n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 82 | 72
percentage of participants
  New onset (n=82,72) | 18.3 | 5.6
  New onset at 1 year (n=82,72) | 14.6 | 2.8
  New onset at 2 years (n=70,70) | 4.3 | 2.9
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; New onset (from baseline up to On-Therapy Month 24); Test type: Superiority or Other; p = 0.025, Fisher Exact — Alpha was unadjusted
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; New onset at 1 year (from baseline up to On-Therapy Month 12); Test type: Superiority or Other; p = 0.012, Fisher Exact — Alpha was unadjusted
Statistical Analysis 3: Comparison: Sirolimus vs Tacrolimus; New onset at 2 years (from On-Therapy Month 12 to On-Therapy Month 24); Test type: Superiority or Other; p = 1.000, Fisher Exact — Alpha was unadjusted

33. Secondary Outcome: Percentage of Participants With New-Onset Diabetes Receiving Treatment for Diabetes (Insulin and Non-Insulin)
Description: Participants were considered as having new onset diabetes during the On-therapy period if any of the below events emerged between baseline and Month 12 or Month 24: 1) at least 30 days continuous, or at least 25 days non-stop (without gap) use of any diabetic treatment after randomization; 2) a fasting glucose ≥126 mg/dL after randomization; or 3) a non-fasting glucose ≥200 mg/dL after randomization.
Time Frame: 12 Months and 24 Months
Population: Safety Population. Only participants with new-onset diabetes mellitus at the beginning of the analysis interval were included; those with pre-existing diabetes were excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 15 | 4
percentage of participants
  Insulin (12-Month) | 13.3 | 0.0
  Insulin (24-Month) | 6.7 | 25.0
  Non-insulin (12-Month) | 13.3 | 0.0
  Non-Insulin (24-Month) | 13.3 | 0.0
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Insulin (12-Month); Test type: Superiority or Other; p = 1.000, Fisher Exact — Alpha was unadjusted
Statistical Analysis 2: Comparison: Sirolimus vs Tacrolimus; Non-insulin (12-Month); Test type: Superiority or Other; p = 1.000, Fisher Exact — Alpha was unadjusted
Statistical Analysis 3: Comparison: Sirolimus vs Tacrolimus; Non-insulin (24-Month); Test type: Superiority or Other; p = 0.386, Fisher Exact — Alpha was unadjusted
Statistical Analysis 4: Comparison: Sirolimus vs Tacrolimus; Insulin (24-Month); Test type: Superiority or Other; p = 1.000, Fisher Exact — Alpha was unadjusted

34. Secondary Outcome: Percentage of Participants With Infection
Description: Includes adverse events based on categorization by the investigator as 'infection', regardless of the event preferred term in MedDRA.
Time Frame: From randomization up to 24 months after transplantation (On-Therapy)
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants | 61.8 | 52.0
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.129, Fisher Exact

35. Secondary Outcome: Percentage of Participants With Cytomegalovirus (CMV) Infection
Description: Includes adverse event terms reported by the investigator to be attributed to the organism 'cytomegalovirus', regardless of the preferred term in MedDRA.
Time Frame: From randomization up to 24 months after transplantation (On-Therapy)
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants | 3.1 | 3.3
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 1.000, Fisher Exact

36. Secondary Outcome: Percentage of Participants With Polyomavirus Infection
Description: Includes adverse event terms reported by the investigator to be attributed to the organism 'polyomavirus', regardless of the preferred term in MedDRA.
Time Frame: From randomization up to 24 months after transplantation (On-Therapy)
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants | 3.8 | 7.3
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.276, Fisher Exact

37. Secondary Outcome: Percentage of Participants With Malignancy
Description: Includes any adverse events based on categorization by the investigator as 'malignancy', regardless of the event preferred term in MedDRA.
Time Frame: From randomization up to 24 months after transplantation (On-Therapy)
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 131 | 123
percentage of participants | 3.1 | 7.3
Statistical Analysis 1: Comparison: Sirolimus vs Tacrolimus; Test type: Superiority or Other; p = 0.158, Fisher Exact

ADVERSE EVENTS:
Time Frame: From randomization up to 24 months after transplantation (plus [+]4 weeks) for adverse events (AEs) and serious AEs (SAEs).
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sirolimus | Tacrolimus
Serious Adverse Events (participants affected / at risk) | 50/131 | 38/123
Other Adverse Events (participants affected / at risk) | 116/131 | 88/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=131) | Tacrolimus (N=123)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1
Gingivitis ulcerative (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Granuloma (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Pseudopolyp (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 1
Sudden cardiac death (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Kidney transplant rejection (Immune system disorders) | 3 | 1
Transplant rejection (Immune system disorders) | 11 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Ateriovenous fistula site infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Osteomyelitis bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 3
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia cryptococcal (Infections and infestations) | 1 | 0
Polyomavirus-associated nephropathy (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respriatory tract infection (Infections and infestations) | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 5 | 2
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Immunosuppressant drug level increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Thalamic infarction (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 3 | 0
Renal cyst ruptured (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 2
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=131) | Tacrolimus (N=123)
Leukopenia (Blood and lymphatic system disorders) | 11 | 9
Polycythaemia (Blood and lymphatic system disorders) | 2 | 7
Apthous stomatitis (Gastrointestinal disorders) | 13 | 1
Diarrhoea (Gastrointestinal disorders) | 22 | 12
Mouth ulceration (Gastrointestinal disorders) | 16 | 0
Nausea (Gastrointestinal disorders) | 7 | 9
Stomatitis (Gastrointestinal disorders) | 11 | 1
Vomiting (Gastrointestinal disorders) | 4 | 7
Oedema peripheral (General disorders) | 25 | 9
Pyrexia (General disorders) | 13 | 6
Nasopharyngitis (Infections and infestations) | 7 | 6
Upper respiratory tract infection (Infections and infestations) | 22 | 13
Urinary tract infection (Infections and infestations) | 14 | 8
Blood creatinine increased (Investigations) | 8 | 5
Weight increased (Investigations) | 7 | 4
Dyslipidemia (Metabolism and nutrition disorders) | 15 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 14 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 9
Headache (Nervous system disorders) | 16 | 7
Tremor (Nervous system disorders) | 0 | 8
Proteinuria (Renal and urinary disorders) | 19 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Acne (Skin and subcutaneous tissue disorders) | 19 | 1
Hypertension (Vascular disorders) | 11 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.